CLINICAL TRIAL: NCT04993196
Title: Quantitative T1rho Magnetic Resonance Imaging in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Tiffany So, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TSo
Record Dates: First submitted 2021-07-26; First posted 2021-08-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T1rho MRI (Experimental)
  Interventions: Diagnostic Test: T1rho imaging

INTERVENTIONS:
Diagnostic Test: T1rho imaging — Magnetic Resonance Imaging using T1rho

SUMMARY:
T1rho imaging is a new MRI technique that has strong potential in neuroimaging. This technique does not require exogenous contrast agents and has high spatial resolution.

In this study we aim to characterise the normal appearance of T1rho in the brain parenchyma in healthy participants. T1rho values will be measured in normal brain structures.

ELIGIBILITY:
Inclusion Criteria:

- Male and female volunteers greater than or equal to 18 years of age

Exclusion Criteria:

* Subjects with a contraindication to magnetic resonance imaging such as the presence of metallic implants, claustrophobia and pregnancy.
* Subjects with previous severe allergic or anaphylactoid reaction to a gadolinium contrast agent, or contraindication to contrast gadolinium administration, such severe renal disease or acutely deteriorating renal function, who would be at risk of nephrogenic systemic fibrosis
* Subjects who are unable to tolerate the scan without moving the head as a result of symptoms such as tremor, spasticity, involuntary movements and spasms, cognitive impairment, coughing, and shortness of breath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
T1rho value in normal grey and white matter in healthy volunteers | Up to 2 months
  T1rho value (measured on T1rho weighted MRI) in normal grey and white matter in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No